CLINICAL TRIAL: NCT00003795
Title: Quality of Life of Gynecologic Cancer Survivors
Brief Title: Quality of Life in Survivors of Gynecologic Cancer
Status: Completed | Type: Observational
Sponsor: Gynecologic Oncology Group (Network)
Collaborators: National Cancer Institute (NCI) (NIH)
Organization: GOG Foundation (Network)
Other Study IDs: CDR0000066938; GOG-9902
Record Dates: First submitted 1999-11-01; First posted 2003-07-18 (Estimated); Last update posted 2013-05-27 (Estimated); Status verified 2009-03

CONDITIONS: Endometrial Cancer; Ovarian Cancer
Keywords: stage I ovarian epithelial cancer; stage II ovarian epithelial cancer; stage I endometrial carcinoma; stage II endometrial carcinoma
MeSH Terms: conditions — Endometrial Neoplasms; Ovarian Neoplasms; Carcinoma, Ovarian Epithelial

INTERVENTIONS:
Procedure: quality-of-life assessment

SUMMARY:
RATIONALE: Quality-of-life assessment in cancer survivors may help determine the long-term effects of having had gynecologic cancer and may help improve the quality of life for future cancer survivors.

PURPOSE: This clinical trial is studying the quality of life in survivors of gynecologic cancer.

DETAILED DESCRIPTION:
OBJECTIVES:

* Describe the significant quality of life (QOL) concerns and long term survivorship issues of women diagnosed and treated for early stage ovarian and endometrial cancer five or more years ago.
* Identify mechanisms which contribute to a gynecologic cancer survivorship model through comparison and prediction of high versus low QOL associated with long term adjustment and survivorship. Examine social support, coping efforts, self-efficacy, meaning associated with survivorship, performance status, and age at diagnosis as potential predictors.
* Identify and compare factors that predict high versus low QOL for women with early stage endometrial cancer completing participation in GOG-99 clinical trial. Conduct exploratory analysis examining long term QOL concerns of survivors randomized to surgery arm with or without radiotherapy.

OUTLINE: Patients complete one telephone interview with a professional female interviewer. The interview lasts approximately 60 minutes and is audiotaped.

PROJECTED ACCRUAL: A total of 197 early stage endometrial cancer survivors and 114 early stage ovarian cancer survivors will be accrued for this study within 2 years.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically confirmed early stage ovarian and endometrial cancer survivors treated and diagnosed five or more years ago
* Patients completing treatment in GOG-95 or GOG-99 protocols at least 5 years ago with no recurrence of disease
* Patients with secondary malignancy or under treatment for other medical conditions are eligible

PATIENT CHARACTERISTICS:

Age:

* Not specified

Performance status:

* Not specified

Life expectancy:

* Not specified

Hematopoietic:

* Not specified

Hepatic:

* Not specified

Renal:

* Not specified

Other:

* Must be capable of completing telephone interview in English

PRIOR CONCURRENT THERAPY:

Biologic therapy:

* See Disease Characteristics

Chemotherapy:

* See Disease Characteristics

Endocrine therapy:

* See Disease Characteristics

Radiotherapy:

* See Disease Characteristics

Surgery:

* See Disease Characteristics

Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 311 (Estimated)
Dates: Start 1999-04; Primary Completion 2002-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Lari B. Wenzel, PhD, Study Chair — Chao Family Comprehensive Cancer Center
Locations (44):
- United States (43):
  - University of Alabama at Birmingham Comprehensive Cancer Center, Birmingham, Alabama
  - Jonsson Comprehensive Cancer Center, UCLA, Los Angeles, California
  - Community Hospital of Los Gatos, Los Gatos, California
  - Chao Family Comprehensive Cancer Center, Orange, California
  - University of Colorado Cancer Center, Denver, Colorado
  - Walter Reed Army Medical Center, Washington D.C., District of Columbia
  - H. Lee Moffitt Cancer Center and Research Institute, Tampa, Florida
  - Rush-Presbyterian-St. Luke's Medical Center, Chicago, Illinois
  - University of Chicago Cancer Research Center, Chicago, Illinois
  - Indiana University Cancer Center, Indianapolis, Indiana
  - Holden Comprehensive Cancer Center at The University of Iowa, Iowa City, Iowa
  - Albert B. Chandler Medical Center, University of Kentucky, Lexington, Kentucky
  - New England Medical Center Hospital, Boston, Massachusetts
  - University of Massachusetts Memorial Medical Center, Worcester, Massachusetts
  - University of Mississippi Medical Center, Jackson, Mississippi
  - Washington University School of Medicine, St Louis, Missouri
  - CCOP - Montana Cancer Consortium, Billings, Montana
  - Cooper Hospital/University Medical Center, Camden, New Jersey
  - Cancer Center of Albany Medical Center, Albany, New York
  - State University of New York Health Science Center at Brooklyn, Brooklyn, New York
  - Schneider Children's Hospital at North Shore, Manhasset, New York
  - Memorial Sloan-Kettering Cancer Center, New York, New York
  - University of Rochester Cancer Center, Rochester, New York
  - State University of New York Health Sciences Center - Stony Brook, Stony Brook, New York
  - Lineberger Comprehensive Cancer Center, UNC, Chapel Hill, North Carolina
  - Duke Comprehensive Cancer Center, Durham, North Carolina
  - Comprehensive Cancer Center at Wake Forest University, Winston-Salem, North Carolina
  - Barrett Cancer Center, The University Hospital, Cincinnati, Ohio
  - Ireland Cancer Center, Cleveland, Ohio
  - Cleveland Clinic Taussig Cancer Center, Cleveland, Ohio
  - Arthur G. James Cancer Hospital - Ohio State University, Columbus, Ohio
  - University of Oklahoma College of Medicine, Oklahoma City, Oklahoma
  - Abington Memorial Hospital, Abington, Pennsylvania
  - Milton S. Hershey Medical Center, Hershey, Pennsylvania
  - University of Pennsylvania Cancer Center, Philadelphia, Pennsylvania
  - Kimmel Cancer Center of Thomas Jefferson University - Philadelphia, Philadelphia, Pennsylvania
  - Fox Chase Cancer Center, Philadelphia, Pennsylvania
  - Medical University of South Carolina, Charleston, South Carolina
  - Brookview Research, Inc., Nashville, Tennessee
  - Simmons Cancer Center - Dallas, Dallas, Texas
  - University of Texas - MD Anderson Cancer Center, Houston, Texas
  - Fred Hutchinson Cancer Research Center, Seattle, Washington
  - Tacoma General Hospital, Tacoma, Washington
- Tom Baker Cancer Center - Calgary, Calgary, Alberta, Canada